CLINICAL TRIAL: NCT03852342
Title: Reactive Doses and Times During Oral Food Challenge (OFC) to Peanut
Brief Title: Reactive Doses and Times During Oral Food Challenge to Peanut
Acronym: PeaNewT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0344
Record Dates: First submitted 2018-09-12; First posted 2019-02-25 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Peanut Allergy
Keywords: Anaphylaxis; Oral Food Challenge; Hypersensitivity; Food Allergy; Peanut
MeSH Terms: conditions — Peanut Hypersensitivity; Anaphylaxis; Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peanut allergy is a growing public health problem in developed countries with more and more hospitalizations for anaphylaxis. It has been determined that sensitization to certain peanut proteins such as rAra h 2, is predictive of allergy and could predict the severity of reaction (anaphylaxis) during Oral food challenges (OFC). So far, consensual threshold for cutaneous test and IgE as predictor in the positivity of OFC have not been determined. Identification of reactive doses for OFC and phenotype of patients would help to personalize management of patients subgroups, with an optimal security.

ELIGIBILITY:
Inclusion criteria:

* Patients with a clinical suspicion of peanut allergy who underwent OFC to peanut
* Patients not objecting to participate in the study
* Men and women are included

Exclusion criteria:

• The patient refused to participate in the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a clinical suspicion of peanut allergy who underwent an open OFC to peanut between June 2001 to July 2018 in the Allergy Unit of the University Hospital of Montpellier (France).
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Reactive doses of peanut (mg) at which an allergic reaction appears in patients with positive peanut Oral Food Challenge | 1 day
  An Oral Food Challenge consists in the ingestion of the suspected allergic food. The patient is given increased dose levels of this food throughout a day. The OFC is positive when the patient presents a clinical reaction (clinical symptoms linked to an allergic response) triggered by the food ingested.
  We'll gather the data of all patients who came in our unit of Allergology and who had a positive peanut OFC.
  The reactive dose is calculated from the total cumulative dose (mg) of peanut reached when the OFC peanut is considered positive.
  The reactive dose is considered as a time dependent data and will be analyzed with survival data analysis methods.
  The analyzed event is a positive OFC

SECONDARY OUTCOMES:
Time between the reaction and the last administered dose | 1 day
  Time between the reaction and the last administered dose
Identifying risk factors of peanut hypersensitivity | 1 day
  To identify the risk factors, that remain significantly associated with a positive peanut OFC
Risk factors of anaphylaxis during a positive peanut OFC | 1 day
  To identify, among the collected data on the patient's clinical history detailled below, the risk factors of occurrence of an anaphylactic reaction during peanut OFC.
  Anaphylaxis is defined as a severe allergic reaction that appears quickly and has a fatal potential. It is usually characterized by the appearance of several signs and symptoms that can affect one or more systems of our body.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEMOLY, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No